CLINICAL TRIAL: NCT06598709
Title: International Survey for EXTubation Evaluation and Respiratory Dynamics in Acute Respiratory Distress Syndrome
Acronym: EXTEND ARDS
Status: Enrolling by invitation | Type: Observational
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Mitsuaki Nishikimi, Assistant Professor Department of Emergency and Critical Care Medicine, Graduate School of Biomedical and Health Sciences, Hiroshima University, Hiroshima University
Other Study IDs: EXTEND_ARDS_study; EXTEND_ARDS_study (Registry Identifier: EXTEND_ARDS_study)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome)
Keywords: extubation; ARDS; SBT; Spontaneous Breathing Trial; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mechanically ventilated adult ARDS patients: Adult mechanically ventilated patients (≥ 16 years old) expected to receive invasive mechanical ventilator for more than 48 hours

SUMMARY:
EXTEND ARDS study is an international survey for ventilator weaning and extubation among ARDS patients. This study will be conducted on behalf of the Japanese ARDS Clinical Practice Guideline 2024 Committee as well as endorsement of the Japanese Society of Intensive Care Medicine, the Japanese Respiratory Society, and the Japanese Society of Respiratory Care Medicine. This survey aims to prospectively collect the clinical data of mechanically ventilated ARDS patients related with ventilator weaning and extubation internationally as well as the outcome of ARDS patients with extubation failure. This study also aims to identify predictive factors strongly associated with extubation failure. The contents of mechanical ventilation settings, respiratory conditions, and blood examination data will be collected.

DETAILED DESCRIPTION:
1.1. Background

Acute respiratory distress syndrome (ARDS) is a life-threatening condition characterized by widespread inflammatory lung injury, and is encountered in an estimated 23% of mechanically ventilated patients (1). Recent studies reported that the mortality of mechanically ventilated patients with ARDS was still as high as approximately 40% (1), which implies that better management strategies for them are needed to improve the outcomes.

In the management for the mechanical ventilated patients with ARDS, the timing and judgement for extubation is clinically important, because extubation failure can be associated with worse outcome (2). The most recent ARDS guidelines recommend a weaning protocol for extubation and introduced several predictive clinical factors for extubation failure, but they are mainly based on the studies for patients with acute respiratory failure (3), and there is no study focusing on the patients with ARDS. Considering that the best method to extubate successfully has not been determined, the clinical management at the timing of extubation can be varied by each institution or each country, and the investigators thought that international survey focusing on the management for extubation of ARDS patients would be needed.

1.2. Significance of the study

Our international survey can identify the management associated with better outcome as well as clinical factors to predict extubation failure at the timing of extubation attempt. This study will contribute to the development of better management for extubation and thereby improve the outcomes of patients with ARDS.

This study has the potential to increase the generalizability of the results which will be obtained from all regions of the world, including Asia, Europe, North and South America, Oceania, and Africa. Therefore, the results will potentially contribute to improving patient outcomes in all regions of the world. Furthermore, the results obtained will provide a detailed picture of the current ICU management given to mechanical ventilated patients with ARDS in the ICU.

1.3．Study Design

This study is international multicenter prospective survey.

2. Aim of the study and evaluation items 2.1. Study Hypothesis

* Mortality of ARDS patients with extubation failure is higher than those without failure.
* Management and timing for ventilator weaning and extubation failure is different by each institution, each country, or each continent, some of which is associated with their outcome.
* Some clinical factors for predicting extubation failure is identified.

2.2. Aim of the study Aim 1: Describing epidemiology, management, timing, and outcome for ventilator weaning and extubation of ARDS patients in the world Aim 2: Comparing the protocol for weaning and extubation between the ARDS patients who had successful extubation and those who did not Aim 3: Comparing the change of respiratory mechanics in the SBT and post-extubation between the ARDS patients who had successful extubation and those who did not Aim 4: Identifying clinical factor available during SBT and in the early times after extubation for predicting extubation failure

ELIGIBILITY:
Inclusion Criteria:

1. Adult mechanically ventilated patients (≥ 16 years old) expected to receive invasive mechanical ventilator for more than 48 hours
2. Patients who meet the diagnosis of ARDS at the start of invasive mechanical ventilation based on a new global definition of ARDS.

Exclusion Criteria:

1. Patients who already had tracheostomy at the start of invasive mechanical ventilation
2. Patients who were transferred to participating hospital more than 2 days after the start of invasive mechanical ventilation
3. Patients with terminal conditions at the start of invasive mechanical ventilation
4. Patients who have expressed their refusal to have their clinical data used in research

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult mechanically ventilated patients (≥ 16 years old) expected to receive invasive mechanical ventilator for more than 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
90 days in-hospital mortality | From intubation to 90 days after intubation
  90 days in-hospital mortality
occurrence of re-intubation event | From extubation until the hospital discharge, assessed up to 24 months
  occurrence of re-intubation event

CONTACTS AND LOCATIONS:
Locations (1):
- Hiroshima university hospital, Hiroshima, Japan

IPD SHARING:
Plan to Share IPD: Yes
Study protocol